CLINICAL TRIAL: NCT01033474
Title: Embryonic Developmental Rates and Pregnancies Following the Vitrification of Human Oocytes Using Two Methodologies.
Brief Title: Results Following the Vitrification of Human Oocytes Using 2 Methodologies
Status: Withdrawn | Type: Observational
Why Stopped: NW Center for Reproductive Sciences was sold and is no longer open
Sponsor: Northwest Center for Reproductive Sciences (Other)
Responsible Party: Klaus Wiemer PhD, Pranor and NW Center for Reproductive Sciences
Other Study IDs: 555-2009
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Infertility
Keywords: Infertile Patients
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- donor eggs
- infertile patients

SUMMARY:
The investigators are going to compare embryo developmental rates of human eggs following freezing in two different freezing methods. The investigators are going to compare the pregnancy rates following transfer to patients as well.

Null Hypothesis: The type of vitrification methodology used will not have an impact on the following:

* Survival rates
* Embryonic developmental rates
* Pregnancy and implantation rates.

DETAILED DESCRIPTION:
Randomization of Oocytes: Oocytes will be denuded approximately 1-2 hours post retrieval and graded for maturity. Only the Metaphase II oocyte will be vitrified. Half of the oocytes within each donor will be randomized to the following treatments.

1. Frozen using an open system using a metal grid to hold the oocyte. Three to five oocytes will be frozen on the metal grid using a minute amount (< 2-3 µls) of cryoprotectant. A top is put over the metal grid to protect the oocytes. This system has proven to be successful in limited cases in Peru. This is an open system of vitrification where the oocytes are directly plunged into liquid nitrogen. This will serve as the control.
2. Frozen in closed straws using a methodology developed by Jim Stachecki. Three to five oocytes will be frozen in ¼ cc straws. This is very similar to the method used to successfully vitrify blastocysts. This will be the experimental treatment.

Null Hypothesis: The type of vitrification methodology used will not have an impact on the following:

* Survival rates
* Embryonic developmental rates
* Pregnancy and implantation rates. Measured Outcomes The effect of vitrification technique will be measured using the appropriate statistical analysis on the following parameters.

  1. Survival rates following thawing.
  2. Effect of vitrification technique on how oocytes react to ICSI. The parameters have been previously defined at NCRS.
  3. Normal fertilization rates, abnormal fertilization rates and rates of degeneration following ICSI.
  4. Embryonic development rates. Embryos will be cultured until Day 5/6 and rate as well as quality of blastocyst will be noted.
  5. Pregnancy and implantation rates following replacement in endometrial prepared recipients.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy and pass testing as per clinic standards

Exclusion Criteria:

* Are over the age or cannot carry a pregnancy safely

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will use infertile patients that need donor oocytes
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-09 (Estimated); Study Completion 2011-07 (Actual)

SECONDARY OUTCOMES:
Pregnancy rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorio de Reproducción Asistida, Lima, Peru